CLINICAL TRIAL: NCT05615818
Title: Molecular Targeted Maintenance Therapy Versus Standard of Care in Advanced Biliary Cancer: an International, Randomised, Controlled, Open-label, Platform Phase 3 Trial
Brief Title: Personalized Medicine for Advanced Biliary Cancer Patients
Acronym: SAFIR-ABC10
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Cancer Research UK & UCL Cancer Trials Centre (Other); Belgian Group of Digestive Oncology (Other); National Cancer Institute, France (Other Government); Cancer Research UK (Other); Taiho Oncology, Inc. (Industry); Servier (Industry); Zymeworks BC Inc. (Industry); Accord Healthcare, Inc. (Industry); Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-GMP-2201 - PRODIGE 78; 2022-000190-19 (EudraCT Number); 2022-502403-30-00 (Other: EU-CT)
Record Dates: First submitted 2022-10-28; First posted 2022-11-14 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2024-11

CONDITIONS: Biliary Tract Neoplasms
Keywords: Biliary Tract Neoplasms; Targeted therapy; Personalised medicine
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — futibatinib; ivosidenib; zanidatamab; Trastuzumab; neratinib; encorafenib; binimetinib; niraparib; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Molecular targeted therapy matched to genetic alteration carried by the tumour
  Interventions: Drug: Futibatinib; Drug: Ivosidenib; Drug: Zanidatamab; Drug: Trastuzumab; Drug: Neratinib; Drug: Encorafenib; Drug: Binimetinib; Drug: Niraparib
- Control (Active Comparator): Continued standard of care treatment for first-line biliary tract cancer
  Interventions: Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Futibatinib — Dose 20 mg once a day (QD)
  Arms: Experimental
Drug: Ivosidenib — Dose 500 mg QD
  Other Names: Tibsovo
  Arms: Experimental
Drug: Zanidatamab — Dose: Patients < 70 kg: 1800 mg every 3 weeks (Q3W), Patients ≥ 70 kg: 2400 mg Q3W
  Arms: Experimental
Drug: Trastuzumab — Loading dose 8 mg/kg, then 6 mg/kg Q3W (Combination with neratinib)
  Other Names: Zercepac
  Arms: Experimental
Drug: Neratinib — Dose: 240 mg QD (combination with trastuzumab)
  Other Names: Nerlynx
  Arms: Experimental
Drug: Encorafenib — Dose: 450 mg QD (Combination with binimetinib)
  Other Names: Braftovi
  Arms: Experimental
Drug: Binimetinib — Dose: 45 mg twice a day (BID) (Combination with encorafenib)
  Other Names: Mektovi
  Arms: Experimental
Drug: Niraparib — Dose: 200 mg QD or 300 mg QD
  Other Names: Zejula
  Arms: Experimental
Drug: Cisplatin — Dose: 25 mg/m2 IV on days 1 and 8 Q3W (CISGEM)
  Arms: Control
Drug: Gemcitabine — Dose: 1000 mg/m2 IV on days 1 and 8 Q3W (CISGEM)
  Arms: Control

SUMMARY:
The object of this trial is to evaluate whether the introduction of a targeted therapy after 4 cycles of the current standard-of-care treatment for advanced biliary cancer is superior to continuing with the standard treatment.

The trial is composed of two phases: (i) An initial screening phase to identify a suitable patient population, during which a molecular profile of the patient's tumour will be obtained, and (ii) a randomised comparative trial in which patients with disease control after 4 cycles of standard treatment, and whose tumour harbours a targetable molecular alteration, will be randomised (2:1) to receive either a matched targeted therapy or to continue with the standard treatment.

DETAILED DESCRIPTION:
This is a Phase 3, multicentre, randomised, open-label trial to evaluate whether the introduction of molecular targeted therapy (MTT) as maintenance after 4 cycles of standard-of-care first-line systemic therapy (1L SoC) is superior to continuation of 1L-SoC in the treatment of patients with ABC. The trial is composed of two phases: (i) An initial screening phase to identify a suitable patient population, and (ii) a randomised comparative trial.

The aim of the screening phase is to identify a medically suitable population, to obtain a molecular profile of the patient's tumour, to collect baseline data concerning patient demographics and disease characteristics and to obtain pre-treatment blood and tumour samples for further translational research.

A genetic profile will be obtained from tumour-derived DNA and RNA samples by next-generation sequencing and from circulating tumour DNA. The trial Molecular Tumour Board will determine whether each patient harbours a targetable molecular alteration for one or more of the trial MTTs.

Patients with disease control after 4 cycles of 1L-SoC, who did not experience limiting toxicity, and whose tumour harbours at least one targetable molecular alteration, will be invited to participate in the randomised phase of the trial in which 159 eligible patients will be randomised (2:1) to receive either maintenance therapy with a matched MTT or to continue 1L-SoC treatment.

ELIGIBILITY:
SCREENING PHASE

Inclusion Criteria:

1. Signed a written informed consent form prior to any trial specific procedures (Consent #1)
2. Histologically-proven intrahepatic, perihilar or distal cholangiocarcinoma, or gallbladder carcinoma (ampullary carcinoma excluded)
3. De novo or recurrent, locally advanced (non-resectable) or metastatic disease
4. Availability of a suitable archived sample of primary or metastatic tumour tissue (frozen, or FFPE) or able to undergo a biopsy to obtain a suitable malignant tissue sample
5. Aged ≥18 years
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Estimated life expectancy >3 months
8. Candidate for 1L-SoC therapy, or has initiated first cycle of 1L-SoC therapy
9. Affiliated to a social security system or in possession of equivalent private health insurance (according to local country health provision arrangements).

Exclusion Criteria:

1. Contraindication to 1L-SoC
2. Patients who are candidates for locoregional therapy
3. Contraindication to tumour biopsy in the absence of suitable archived sample of tumour tissue
4. Prior anticancer therapy in the palliative setting. Adjuvant capecitabine allowed if completed ≥ 183 days prior to study entry
5. Received more than 1 cycle of treatment with 1L-SoC
6. Prior treatment with any of the MTT under investigation in the SAFIR-ABC10 study
7. Current malignancies (other than ABC), with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for 5 years or more and are deemed at negligible risk for recurrence, are eligible for the trial
8. Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol
9. Women who are pregnant or breast-feeding
10. Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons
11. Individuals deprived of liberty or placed under protective custody or guardianship

RANDOMISED TRIAL

Inclusion Criteria:

1. Signed a written informed consent form prior to any trial specific procedures (Consent #2)
2. Molecular profile showing the tumour harbours at least one targetable molecular alteration with a MTT in the study portfolio (as determined by the trial MTB)
3. Disease control (stable or responsive) after 4 cycles of 1L-SoC, compared to a pre-treatment disease evaluation, as assessed by the investigator
4. ECOG performance status of 0 or 1
5. Presence of at least one evaluable lesion according to RECIST v1.1, or complete response to 12 weeks 1L-SoC
6. Adequate bone marrow function: absolute neutrophil count (ANC) ≥1.5 × 10⁹/L, platelet count ≥100 × 10⁹/L, and haemoglobin ≥9 g/dL
7. Adequate liver function: total bilirubin level ≤1.5 × the upper limit of normal (ULN) range (total bilirubin ≤3.0 ULN when the patient has documented Gilbert syndrome), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤2.5 × ULN (AST and ALT ≤5 ULN when documented tumour liver involvement)
8. Adequate renal function: estimated creatinine clearance ≥ 60 mL/min according to the Cockcroft-Gault formula
9. Adequate cardiac function: left ventricular ejection fraction ≥50% at baseline as determined by either echocardiogram or multigated acquisition scan (MUGA)
10. Adequate biliary drainage, with no evidence of ongoing infection
11. Men, and women of childbearing potential (WOCBP) must agree to use adequate contraception for the duration of trial participation and as required after completing study treatment. Men must also agree to not donate sperm and women must agree to not donate oocytes during the specified period.
12. Women of childbearing potential must have a negative serum pregnancy test performed within 3 days before the date of randomisation
13. Willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan, laboratory tests, and other study procedures
14. Affiliated to a social security system or in possession of equivalent private health insurance (according to local country health provision arrangements)

Exclusion Criteria:

1. Disease progression occurring at any time prior randomisation, or toxicity that led to the discontinuation of the 1L-SoC before 4 full cycles have been delivered
2. Toxicities from 1L-SoC not resolved to Grade ≤ 1 (according to version 5.0 the National Cancer Institute - Common terminology criteria for adverse events [NCI-CTCAE v5.0]) before randomisation, with the exception of alopecia
3. Contraindication or known hypersensitivity to the MTT for the molecular alteration found in the patient, or any component in their formulation Note: For patients with multiple target alterations, contraindication to one MTT will not warrant exclusion if MTT to an alternative target is feasible.
4. Microsatellite instability high (MSI-H) or mismatch repair deficient (dMMR) cancers
5. Major surgery within 4 weeks of randomisation
6. Radiotherapy within 7 days of randomisation
7. Untreated central nervous system (CNS) metastases, symptomatic CNS metastases, or radiation treatment for CNS metastases within 4 weeks of start of study treatment. Stable, treated brain metastases are allowed (defined as subjects who are off steroids and anticonvulsants and are neurologically stable with no evidence of radiographic progression for at least 4 weeks at the time of screening).
8. Clinically significant cardiovascular disease (recent acute myocardial infarction, treated congestive heart failure [2 or above on the New York Heart Association functional classification scale], recent thromboembolic or cerebrovascular events [within 12 weeks, excepted if related to indwelling catheter], known prolonged QT syndrome).
9. Cardiorespiratory pathologies where hyperhydration is contraindicated.
10. Manifestation of tinnitus and/or hearing loss since initiation of cisplatin therapy.
11. Known leptomeningeal disease. If leptomeningeal disease has been reported radiographically on baseline magnetic responance imaging (MRI), but is not suspected clinically by the investigator, the subject must be free of neurological symptoms.
12. Concurrent malignancy (other than ABC), with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for 5 years or more and are deemed at negligible risk for recurrence, are eligible for the trial
13. Concomitant treatment with phenytoin in prophylactic use where this cannot be substituted for another therapy
14. Known active hepatitis B virus or hepatitis C virus infection or human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome
15. Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol
16. Women who are pregnant or breast-feeding
17. Participation in another therapeutic trial within the 30 days prior to entering the study. Participation in an observational trial would be acceptable
18. Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons
19. Individuals deprived of liberty or placed under protective custody or guardianship

ADDITIONAL EXCLUSION CRITERIA FOR SPECIFIC MTTs:

Patients assigned to receive oral therapies:

1. Inability or unwillingness to swallow pills
2. History of malabsorption syndrome or other condition that would interfere with enteral absorption. For example, active intestine inflammation (e.g., Crohn's disease or ulcerative colitis) requiring immunosuppressive therapy

Futibatinib:

1. History and/or current evidence of any of the following disorders:

   1. Non-tumour related alteration of the calcium-phosphorus homeostasis that is considered clinically significant in the opinion of the Investigator
   2. Ectopic mineralization/calcification, including but not limited to soft tissue, kidneys, intestine, or myocardia and lung, considered clinically significant in the opinion of the Investigator
   3. Retinal or corneal disorder confirmed by retinal/corneal examination and considered clinically significant in the opinion of the Investigator
2. Concomitant treatment with strong CYP3A/P-gp inhibitors or strong or moderate CYP3A/P gp inducers where these cannot be substituted for another therapy.

Ivosidenib:

1. Patients with history of torsade de pointes
2. Concomitant treatment with digoxin where this cannot be substituted for another therapy
3. Patients with a heart-rate corrected QT interval (using Fridericia's formula) (QTcF) ≥ 450 msec or other factors that increased the risk of QT prolongation or arrhythmic events (e.g. heart failure, hypokalemia, family history of long QT interval syndrome)
4. Concomitant treatment with strong CYP3A4 inducers or dabigatran where these cannot be substituted for another therapy
5. Concomitant treatment with medicinal products known to prolong the QTc interval, or moderate or strong CYP3A4 inhibitors where these cannot be substituted for another therapy
6. Familial history of sudden death or polymorphic ventricular arrhythmia.
7. Hypokalemia, hypomagnesemia or hypocalcemia where this cannot be corrected by supplementation

Zanidatamab:

1. Treatment with anthracyclines within 90 days before first dose of zanidatamab and/or total lifetime load exceeding 360 mg/m2 Adriamycin® or equivalent
2. Use of corticosteroids administered at doses equivalent to > 15 mg per day of prednisone within 2 weeks of first zanidatamab dosing unless otherwise approved by the coordinating investigator. Topical, ocular, intra-articular, intranasal, and/or inhalational corticosteroids are permitted
3. QTcF > 470 ms
4. History of myocardial infarction or unstable angina within 6 months prior to enrollment, troponin levels consistent with myocardial infarction, or clinically significant cardiac disease, such as ventricular arrhythmia requiring therapy, uncontrolled hypertension, or any history of symptomatic congestive heart failure
5. Acute or chronic uncontrolled pancreatitis or Child-Pugh Class C liver disease
6. Clinically significant infiltrative pulmonary disease not related to lung metastases
7. A history of life-threatening hypersensitivity to monoclonal antibodies or recombinant proteins

Neratinib & trastuzumab:

1. Patients with severe hepatic impairment (Child-Pugh Class C)
2. Co-administration with the following medical products that are strong inducers of the CYP3A4/P-gp isoform of cytochrome P450, such as carbamazepine, phenytoin (antiepileptics), St John's wort (Hypericum perforatum) or rifampicin (antimycobacterial)
3. Patients who are experiencing dyspnoea at rest due to complications of advanced malignancy or co-morbidities
4. Hypersensitivity to murine proteins
5. Current active pneumonitis within 90 days of receiving trastuzumab or a known history of interstitial lung disease

Encorafenib & binimetinib:

1. Patients with a history or current evidence of retinal vein occlusion or risk factors for retinal vein occlusion (e.g., uncontrolled glaucoma or history of hyperviscosity or hypercoagulability syndrome)
2. Patients with concurrent neuromuscular disorders associated with elevated creatine phosphokinase (>ULN)
3. Patients with hypokalemia, hypomagnesemia, or hypocalcemia (i.e. Serum potassium, magnesium or calcium < lower normal limit)
4. Patients with a QTcF ≥ 450 msec for men, or ≥ 470 msec for women
5. Current or expected use of a strong inhibitor of CYP3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomisation to disease progression or death, up to 5 years.
  Time from randomisation to the first documented progression of disease (PD) as assessed by the investigator according to RECIST v1.1, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomisation to death, up to 5 years.
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive.
Objective response rate | From randomisation, up to 5 years.
  Objective response rate is defined as the proportion of patients achieving complete response (CR) or partial response (PR) (according to RECIST v1.1). Objective response rate will be presented as the best response achieved compared to the disease assessment performed at randomisation.
Time to treatment failure | From randomisation to treatment failure event, up to 5 years.
  Time from patient starting their allocated treatment to the date at which a patient first experiences a treatment failure event. The following will be considered as treatment failure events: early treatment discontinuation (regardless of reason), disease progression, death, starting a new treatment after completing scheduled treatment, withdrawal from the study due to any reason or loss to follow-up.
Progression-free survival after next line of treatment (PFS2) | From randomisation to second disease progression or death, up to 5 years.
  Time from randomisation to the date of second disease progression or death, whichever occurs first.
Duration of response | From response to disease progression or death, up to 5 years.
  Duration of response is defined as the time from first documented response (compared to baseline measurement taken at randomisation) until the date of disease progression, as assessed by the investigator according to RECIST v1.1, or death from any cause whichever occurs first.
Disease control rate | From randomisation, up to 5 years.
  Disease control rate is defined as the proportion of randomised patients achieving CR, PR, stable disease (SD)/no evidence of disease (NED) as assessed by the investigator according to RECIST v1.1.
Percentage change in tumour size | From randomisation, up to 5 years.
  Taking the measurements at randomisation as the reference.

OTHER OUTCOMES:
Feasibility of molecular screening | Up to 3 months from start of treatment
  The proportion of patients with an available MTB proposition at the time of the 3-month standard of care treatment evaluation.
Quality of life questionnaire - Core 30 (QLQ-C30) | From baseline, every 3 cycles (every 9 weeks) until end of treatment, an average of 1 year
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life Questionnaire - Biliary tract cancer module (QLQ-BIL21) | From baseline, every 3 cycles (every 9 weeks) until end of treatment, an average of 1 year
  This EORTC cholangiocarcinoma and gallbladder cancer specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-BIL21 contains 21 items to assess symptoms. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale.
EuroQOL EQ-5D-5L questionnaire | From baseline, every 3 cycles (every 9 weeks) until end of treatment, an average of 1 year
  Developed by the EuroQol group, the self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials consists of a descriptive system and a visual analogue scale (VAS).
  The EQ-5D-5L descriptive system comprises five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each dimension has 5 levels (1 = "no problems", 2 = "slight problems", 3 = "moderate problems", 4 = "severe problems", and 5 = "extreme problems"). This questionnaire provide a 5-digit score which generate a health state profile. The VAS records the patient's self-rated health on a vertical visual analogue scale where the score range from 0 (The best health you can imagine) to 100 (The worst health you can imagine). The VAS is used as a quantitative measure of health outcome that reflects the patient's own judgement.
Incidence of Adverse Events | From randomisation, up to 5 years
  Safety and tolerability of the treatment will be evaluated using the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5). NCI-CTCAE is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Malka David, MD, Principal Investigator — Institut Mutualiste Montsouris; Julien Edeline, MD, Principal Investigator — Centre Eugène Marquis; Ivan Borbath, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; John Bridgewater, MD, Principal Investigator — University College London Cancer Institute; Juan W Valle, Principal Investigator — University of Manchester and The Christie NHS Foundation Trust
Locations (69):
- Belgium (4):
  - Cliniques universitaires de Bruxelles - Hôpital Erasme ULB, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen (UZA), Edegem
  - Universitair Ziekenhuis Leuven, Leuven
- France (45):
  - CHU Amiens Picardie, Amiens
  - CHU d'Angers, Angers
  - Institut de cancerologie de l'Ouest - Angers, Angers
  - Institut du Cancer Avignon Provence, Avignon
  - CHU de Besançon, Besançon
  - CHU de Bordeaux - Hôpital Haut-Leveque, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU Estaing de Clermont Ferrand, Clermont-Ferrand
  - APHP - Hopital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU Grenoble Alpes, Grenoble
  - Groupe hospitalier mutaliste de Grenoble - Institut Daniel Hollard, Grenoble
  - Centre Oscar Lambret, Lille
  - CHU Lille, Lille
  - CHU Dupuytren, Limoges
  - Centre Leon Bérard, Lyon
  - Clinique Privée Jean Mermoz, Lyon
  - Hospices Civils de Lyon - Croix Rousse, Lyon
  - APHM - CHU La Timone, Marseille
  - Hôpital Européen, Marseille
  - Institut Paoli Calmettes, Marseille
  - Institut de Cancer de Montpellier, Montpellier
  - CHU Nantes - Hôtel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - APHP - Hôpital Beaujon, Paris
  - APHP - Hôpital Cochin, Paris
  - APHP - Hôpital Saint Antoine, Paris
  - Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - Institute Mutualiste Montsouris, Paris
  - CH de Pau, Pau
  - CHU Poitiers, Poitiers
  - CH Cornouaille, Quimper
  - CHU de Reims, Reims
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - CHU Charles Nicolle, Rouen
  - Institut Curie - Saint Cloud, Saint-Cloud
  - Institut de Cancerologie de l'Ouest, Saint-Herblain
  - Hôpital Foch, Suresnes
  - CHU Toulouse, Toulouse
  - CH Valence, Valence
  - CHRU de Nancy, Vandœuvre-lès-Nancy
  - APHP - Hôpital Paul Brousse, Villejuif
  - Gustave Roussy, Villejuif
- United Kingdom (20):
  - Queen Elizabeth Hospital, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Castle Hill Hospital, Cottingham
  - St James's Hospital, Leeds
  - Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Guy's & St Thomas' Hospital, London
  - Hammersmith Hospital, London
  - Royal Free Hospital, London
  - Royal Marsden Hospital, London
  - University College London, London
  - Maidstone Hospital, Maidstone
  - The Christie Hospital, Manchester
  - Mount Vernon Cancer Centre, Northwood
  - Nottingham University Hospital, Nottingham
  - Churchill Hospital, Oxford
  - North West Anglia NHS Foundation Trust, Peterborough
  - Weston Park Cancer Centre, Sheffield
  - Southampton General Hospital, Southampton
  - Singleton Hospital, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.
Access Criteria: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.